CLINICAL TRIAL: NCT03061994
Title: Metabolomic Study of Patients With Cardiomyopathy in China
Brief Title: Metabolomic Study of All-age Cardiomyopathy
Acronym: MAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingIHLBVD2016023
Record Dates: First submitted 2017-02-06; First posted 2017-02-23 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-03

CONDITIONS: Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy; Left Ventricular Non-compaction; Restrictive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathy, Restrictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiomyopathy: Children(older than 18 years old) are diagnosed as cardiomyopathy by three cardiologists and recruited in pediatric heart center,Beijing Anzhen Hospital, recording the results of clinical lab and echocardiography.
  Adults are diagnosed as cardiomyopathy by three cardiologists and recruited in the department of cardiology ,Beijing Anzhen Hospital.
- Control: Healthy children and adults are recruited in Beijing Anzhen Hospital, with negative results of echocardiography and clinical lab examination.

SUMMARY:
This study aims to 1)characterize the differentially expressed metabolites between cardiomyopathy patients and healthy controls,2)identify the specific biomarkers associated with outcomes or risk evaluation in patients with different cardiomyopathies in a follow-up of a cohort and 3)to determine whether differentially expressed may affect the pathological process of cardiomyopathies . Standardized protocols will be used for the assessment of medical history and examinations, laboratory biomarkers, and the collection of blood plasma.

DETAILED DESCRIPTION:
The aim of this study is to analyze metabolomic profile of patients with cardiomyopathy in order to identify biochemical markers with risk stratification and prognostic value. Clinical data of enrolled patients regarding demographics, cardiovascular risk factors，clinical lab data and previous cardiovascular disease will be recorded. Follow up will be at 3 months,6 months,9 months,1 year and 3 years and will be performed by clinical recordings or phone call when necessary. Blood samples of patients with cardiomyopathy are taken when they enrolled. Serum samples will be analyzed by Liquid Chromatograph Mass Spectrometer/Mass Spectrometer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who was diagnosed as cardiomyopathy by medical history, clinical symptoms, laboratory tests including ECG, echocardiography.
2. Subject understands study requirements aand agrees to sign an informed consent form prior to any study procedures

Exclusion Criteria:

1. Endocrine disease known to cause heart muscle disease (including infants of diabetic mothers)
2. History of rheumatic fever
3. Toxic exposures known to cause heart muscle disease (anthracyclines, mediastinal radiation, iron overload or heavy metal exposure)
4. HIV infection or born to an HIV positive mother
5. Kawasaki disease
6. Immunologic disease
7. Uremia, active or chronic
8. Abnormal ventricular size or function that can be attributed to intense 9.physical training or chronic anemia

10.Chronic arrhythmia, unless there are studies documenting inclusion criteria prior to the onset of arrhythmia (except a patient with chronic arrhythmia, subsequently ablated, whose cardiomyopathy persists after two months is not to be excluded) 11.Malignancy 12.Pulmonary parenchymal or vascular disease (e.g., cystic fibrosis, cor pulmonale, or pulmonary hypertension) 13.Ischemic coronary vascular disease 14.Association with drugs (e.g., growth hormone, corticosteroids, cocaine) or other diseases known to cause hypertrophy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A diagnosis of cardiomyopaty is adjudicated by three cardiologists,according to current guidelines when there was clinical evidence of cardiomyopathy together with clinical symptoms of heart failure or echocardiography or imaging evidence.
  age- and gender- mathced healthy controls are also recuitted in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Result of echocardiography | three year
  The whole results of echocardiography report will be recorded. The indicates whi ch can reflect cardiac function including Left ventricular ejection fraction, left ventricular end diastolic diameter, E/A ratio of bicuspid valve will be used to calculate the association with metabolites.

SECONDARY OUTCOMES:
Cardiovascular death | One year/Three year
  The data is collected during follow-up visit at 1/3 years after discharge
Re-hospitalization | One year/Three year
  patients are hospitalized due to heart failure with decreasing left ventricular ejection fraction (LVEF) or worsen symptoms. The data is collected during follow-up visit at 1/3 years after discharge
Heart transplantation | One year/Three year
  patients are hospitalized due to heart failure.The data is collected during follow-up visit at 1/3 years after discharge
malignant arrythmia | One year/Three year
  Ventricular flutter and fibrillation, atrioventricular block,atrial fibrillation or other cardiac arrhythmia leads to syncope or should be Implantable Cardioverter-Defibrillator (ICD) implantation.
Worsening heart failure | These data is collected from the cases' medical record in an average of 1/3/6/9/12/36 months after the sample recruiting
  Worsen heart failure is defined as decreased ejection fraction(left ventricular ejection fraction decreased over 10%), left ventricular ejection fraction <45% and enlarged heart size measured by echocardiography and changing level of New York Heart Association (NYHA) Functional Classification.And patients who undergo left ventricular assist device (LVAD) will also be included.The data is collected during follow-up visit at 3/6/9/12/36 months after enrollment.
Metabolomic profile on Liquid Chromatograph Mass Spectrometer/Mass Spectrometer analysis of plasma sample | The data is collected from lab in an average of 3 month after the sample recruiting
  The results of metabolomics will be measured by mass spectrometry, including lipids, sugars and amino acids. All of metabolites will be quantitative(unit:mol/L). Identification of molecules via Human Metabolites Database will be reported online.

CONTACTS AND LOCATIONS:
Overall Officials: Yulin Li, PhD, Study Director — Beijing Anzhen Hospital Affiliated to Capital Medical University; Yongqiang Lai, MD, Study Director — Beijing Anzhen Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Institute of heart, lung and blood vessel diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No